CLINICAL TRIAL: NCT02952144
Title: Treatment of Dialysis-Related Amyloidosis Using Lixelle® β2-microglobulin Apheresis Column
Brief Title: Post Approval Study of Lixelle for the Treament of Dialysis-Related Amyloidosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaneka Medical America LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KPA-Lixelle-001
Record Dates: First submitted 2016-10-30; First posted 2016-11-02 (Estimated); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Dialysis Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lixelle® treatment (Experimental): 2 years of Lixelle® treatment in the patients with dialysis related amyloidosis (DRA)
  Interventions: Device: Lixelle® treatment
- natural history (No Intervention): 2 years of natural history in the patients with dialysis related amyloidosis (DRA)

INTERVENTIONS:
Device: Lixelle® treatment — The treatment will be performed with the Lixelle® column connected to upstream of the dialyzer in series on the routine HD circuit according to the description in the IFU. The dialyzer and the Kt/V urea in the conventional HD for each patient will be kept equal in Lixelle®-treatment. Since the maximum blood flow rate for Lixelle® is 250 ml/min, the dialysis time will be extended to achieve the target Kt/V urea. The study will not restrict the type of hemodialyzer and other conditions of HD as specified by the physician. However, any changes to the HD procedure should be recorded properly, and the Kt/V urea should be kept equal to that at the enrollment.
  Arms: Lixelle® treatment

SUMMARY:
Dialysis-related amyloidosis (DRA) is a serious complication of long-term hemodialysis (HD). Its pathogenic mechanism involves accumulation of β2-microglobulin (β2M) in the blood. β2M is produced by most cells in the body and is metabolized in the kidney in healthy individuals. However, in HD patients with renal dysfunction, β2M which is not removed entirely by HD accumulates excessively in the blood. Then it forms amyloid fibrils that are deposited in bones, joints, and soft tissues. The fibrils are further modified by advanced glycation end products (AGE), inducing local macrophage infiltration and production of cytokines leading to chronic inflammation and activation of osteoclasts. Consequently, severe complications with various symptoms are developed, which are collectively referred to as DRA.

Lixelle® is a whole-blood β2M apheresis column developed to adsorb and eliminate β2M selectively from the blood of DRA patients. The treatment is performed with Lixelle® connected upstream of the dialyzer in series on a HD circuit in every session. The Lixelle® column contains porous cellulose beads with covalently linked hexadecyl alkyl chain ligands, which selectively adsorb β2M, via a molecular sieving effect because of its porous structure and hydrophobic interaction with ligands. Lixelle® has been used to relieve symptoms and prevent the progression of DRA in Japan since 1996, when health insurance coverage and reimbursement for the treatment were approved by Japanese Ministry of Health, Labor, and Welfare. Improvement of the activities of daily living (ADL) and remission of arthralgia by Lixelle® treatment has been shown in several clinical studies.

DETAILED DESCRIPTION:
In a post-market study on Lixelle® conducted between 1994 and 1997 in Japan, all adverse events in 183 patients (13, 476 treatments) at 58 centers were collected. The most frequent adverse events were temporary hypotension and anemia, which are common in dialysis or any extracorporeal therapy. Since the maximum blood flow rate for Lixelle® is less than the average blood flow rate for the conventional HD in the USA, Lixelle®- treatment requires a longer treatment time to achieve the same Kt/V urea as the conventional HD in the United States. However, the longer dialysis time and the lower blood flow rate are not likely to increase the rate of adverse events. Adverse events (including Serious Adverse Events) will be collected at each treatment whenever they occur and will be analyzed using descriptive statistics.

This is a prospective double-armed study of 2 years of Lixelle®-treatment. The study consists of the study arm of 2 years of Lixelle®-treatment in 30 DRA patients and the natural history arm of 2 years of conventional HD in 10 DRA patients as the descriptive reference.

The primary objective of this study is to assess the safety of Lixelle® in patients in the USA. The secondary objectives of this study are to assess the probable benefit of Lixelle® to increase the β2M reduction rate in a single dialysis session.

Exploratory endpoints are to assess:

1. the changes of DRA symptoms and ADL of the patients treated with Lixelle® using DRAQ (Dialysis-Related Amyloidosis Questionnaire)
2. the changes of QOL of the patients treated with Lixelle® using KDQOL-SF (Kidney Disease Quality of Life Short Form)
3. the pre-treatment β2M levels at baseline, one and two years; and
4. bone cysts at baseline and two years

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving thrice-weekly HD and diagnosed as DRA by one or more of the following 1 to 4 will be included.

  1. Biopsy of any tissue, showing Congo-red positive amyloid fibrils and immunohistochemical stains consistent with β2M
  2. Shoulder ultrasonography showing rotator cuffs greater than 8 mm in thickness, and /or echogenic pads between muscle groups of the rotator cuff
  3. Two or more diagnoses of the following (1) to (5) (1) Polyarthralgia (2) Carpal tunnel syndrome (3) Trigger finger (4) Dialysis-associated spondylosis ((i) or (ii)) (i) Destructive spondyloarthropathy (DSA) (ii) Spinal stenosis (5) Bone cysts (Bone cysts considered to be caused by other diseases such as osteoarthritis, aneurysmal bone cysts and unicameral bone cysts should be excluded.)
  4. Biopsy of any tissue, showing Congo-red positive amyloid fibrils, and one diagnosis or surgical history of criterion 3- (1) to (5)

Exclusion Criteria:

* Patient who meets any of the following 1 to 7 will be excluded from the study.

  1. Patient diagnosed with rheumatoid arthritis
  2. Patient diagnosed with osteoporosis
  3. Patient diagnosed with osteoarthritis
  4. Patient planning to receive renal transplantation during the study
  5. Patient for whom adequate anticoagulation cannot be achieved
  6. Patient for whom extracorporeal circulation therapy is contraindicated, such as those with severe cardiac insufficiency, acute myocardial infarction, severe cardiac arrhythmia, acute seizure disorder, or severe uncontrolled hypertension or hypotension
  7. Patient planning to become pregnant, pregnant, or breast-feeding
  8. Patient unable to understand or answer the questionnaires even with a proper assistance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
the rate of SAE | through 2 years of Lixelle® treatment during the study period
  comparison of incidence of SAE between between the Lixelle® treatment group and the natural history during treatment period (2 years)

SECONDARY OUTCOMES:
β2M reduction rate in Lixelle® treatment (2 year) | comparison between baseline and 2 years (104 weeks) after Lixelle® treatment
  to compare how much blood β2M level have decreased after after Lixelle® treatment against pre-treatment level.
comparison of β2M reduction rate between Lixelle® treatment and natural history | comparison between baseline and 2 years (104 weeks) after Lixelle® treatment
  to compare β2M reduction rate (see Description in Outcome 2) between the Lixelle® treatment grroup and tne natural history group.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Silberzweig, MD, Principal Investigator — The Rogosin Institute
Locations (1):
- The Rogosin Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Argiles A, Mourad G, Kerr PG, Garcia M, Collins B, Demaille JG. Cells surrounding haemodialysis-associated amyloid deposits are mainly macrophages. Nephrol Dial Transplant. 1994;9(6):662-7. doi: 10.1093/ndt/9.6.662. PMID 7970093
- [Background] Inoue H, Saito I, Nakazawa R, Mukaida N, Matsushima K, Azuma N, Suzuki M, Miyasaka N. Expression of inflammatory cytokines and adhesion molecules in haemodialysis-associated amyloidosis. Nephrol Dial Transplant. 1995 Nov;10(11):2077-82. PMID 8643171
- [Background] Chertow GM, Trimbur T, Karlson EW, Lazarus JM, Kay J. Performance characteristics of a dialysis-related amyloidosis questionnaire. J Am Soc Nephrol. 1996 Aug;7(8):1235-40. doi: 10.1681/ASN.V781235. PMID 8866418
- [Background] Carmichael P, Popoola J, John I, Stevens PE, Carmichael AR. Assessment of quality of life in a single centre dialysis population using the KDQOL-SF questionnaire. Qual Life Res. 2000 Mar;9(2):195-205. doi: 10.1023/a:1008933621829. PMID 10983483
- [Background] Kutsuki H. beta(2)-Microglobulin-selective direct hemoperfusion column for the treatment of dialysis-related amyloidosis. Biochim Biophys Acta. 2005 Nov 10;1753(1):141-5. doi: 10.1016/j.bbapap.2005.08.007. Epub 2005 Sep 6. PMID 16168723
- [Result] Gejyo F, Yamada T, Odani S, Nakagawa Y, Arakawa M, Kunitomo T, Kataoka H, Suzuki M, Hirasawa Y, Shirahama T, et al. A new form of amyloid protein associated with chronic hemodialysis was identified as beta 2-microglobulin. Biochem Biophys Res Commun. 1985 Jun 28;129(3):701-6. doi: 10.1016/0006-291x(85)91948-5. PMID 3893430
- [Result] Gejyo F, Odani S, Yamada T, Honma N, Saito H, Suzuki Y, Nakagawa Y, Kobayashi H, Maruyama Y, Hirasawa Y, et al. Beta 2-microglobulin: a new form of amyloid protein associated with chronic hemodialysis. Kidney Int. 1986 Sep;30(3):385-90. doi: 10.1038/ki.1986.196. PMID 3537446
- [Result] Gejyo F, Homma N, Arakawa M. Carpal tunnel syndrome and beta 2-microglobulin-related amyloidosis in chronic hemodialysis patients. Blood Purif. 1988;6(2):125-31. doi: 10.1159/000169494. No abstract available. PMID 3293616
- [Result] Miyata T, Oda O, Inagi R, Iida Y, Araki N, Yamada N, Horiuchi S, Taniguchi N, Maeda K, Kinoshita T. beta 2-Microglobulin modified with advanced glycation end products is a major component of hemodialysis-associated amyloidosis. J Clin Invest. 1993 Sep;92(3):1243-52. doi: 10.1172/JCI116696. PMID 8376584
- [Result] Abe T, Uchita K, Orita H, Kamimura M, Oda M, Hasegawa H, Kobata H, Fukunishi M, Shimazaki M, Abe T, Akizawa T, Ahmad S. Effect of beta(2)-microglobulin adsorption column on dialysis-related amyloidosis. Kidney Int. 2003 Oct;64(4):1522-8. doi: 10.1046/j.1523-1755.2003.00235.x. PMID 12969174
- [Result] Gejyo F, Kawaguchi Y, Hara S, Nakazawa R, Azuma N, Ogawa H, Koda Y, Suzuki M, Kaneda H, Kishimoto H, Oda M, Ei K, Miyazaki R, Maruyama H, Arakawa M, Hara M. Arresting dialysis-related amyloidosis: a prospective multicenter controlled trial of direct hemoperfusion with a beta2-microglobulin adsorption column. Artif Organs. 2004 Apr;28(4):371-80. doi: 10.1111/j.1525-1594.2004.47260.x. PMID 15084199